CLINICAL TRIAL: NCT04749615
Title: Does Periarticular Injection (PAI) Reduce Pain After TKA Among Knee Arthroplasty Patients Receiving Adductor Canal Block and Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee (ACB&IPACK)? A Blinded, Randomized Controlled Trial.
Brief Title: Does PAI Reduce Pain After TKA Among Knee Arthroplasty Patients Receiving ACB & IPACK?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-2096
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-05

CONDITIONS: Total Knee Athroplasty
Keywords: TKA; PAI; ACB; IPACK; Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No PAI + ACB & IPACK (Placebo Comparator): Control: saline injection (same injection technique and volumes as described for the active intervention, of normal saline)
  Interventions: Drug: Saline Control Periarticular Injection (PAI)
- PAI + ACB & IPACK (Active Comparator): Active intervention: Periarticular injection: one deep injection prior to cementation and then a second more superficial injection prior to closure. The deep injection will consist of bupivacaine 0.25% with 1:200,000 epinephrine, 30 cc; morphine, 8 mg/ml, 1cc; methylprednisolone, 40 mg/ml, 1 ml; cefazolin, 500 in 10 ml; normal saline, 22cc. The superficial injection will be 20 ml 0.25% bupivacaine
  Interventions: Drug: Periarticular Injection (PAI)

INTERVENTIONS:
Drug: Periarticular Injection (PAI) — PAI is a widely-utilized, surgeon-performed, analgesic intervention for TKA patients.
  Arms: PAI + ACB & IPACK
Drug: Saline Control Periarticular Injection (PAI) — equal volume of saline will be used in place of analgesics used in PAI injections
  Arms: No PAI + ACB & IPACK

SUMMARY:
The goal of this clinical trial is to determine whether Periarticular Injection (PAI) alongside Adductor Canal Block (ACB) and Infiltration between the Popliteal Artery and Capsule of the Knee (IPACK) block can decrease post-operative pain in patients undergoing primary total knee arthroplasty. The main question it aims to answer is:

• Is ACB/IPACK without PAI as effective as ACB/IPACK with PAI for TKA patients?

Participants will be assigned to one of the following groups at random:

* ACB/PACK with PAI
* ACB/IPACK with saline injection

Participants will also be asked to complete pre- and post-operative questionnaires.

DETAILED DESCRIPTION:
Kim et al (2019) have shown that addition of ACB/IPACK to PAI improves analgesic outcomes (the nerve blocks reduced pain with ambulation and reduced opioid consumption). TKA patients receiving PAI + ACB/IPACK (along with a comprehensive multimodal analgesic program) had low pain scores with ambulation on POD1: 1.7 +/- 1.4 (mean +/- SD, NRS, 0-10 scale). The opioid consumption in the first 24 hours was 40.6 +/- 32.1 (mg oral morphine equivalents).

It is not clear if the PAI component is necessary, given the theoretically nearly complete analgesic effects of the ACB/IPACK block. Additionally, anecdotal evidence indicates that some surgeons at HSS routinely use the PAI and some do not, without obvious large differences in analgesic outcomes. While there may be a 'belt and suspenders' advantage to using PAI in addition to ACB/IPACK, it is not desirable to perform unnecessary procedures.

In this study, we seek to compare the efficacy of ACB/IPACK with and without PAI in TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* Planned use of regional anesthesia
* Ability to follow the major components of the study protocol
* English speaking (Secondary outcomes include questionnaires validated in English only)

Exclusion Criteria:

* Patients younger than 25 years old and older than 80
* Non-English speaking
* Patients intending to receive general anesthesia
* Contraindication to nerve blocks or peri-articular injection
* Patients with an ASA of IV or higher
* Renal insufficiency (ESRD, HD, estimated creatinine clearance < 30 ml/min)
* Patients with major prior ipsilateral open knee surgery
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an Independent review committee ("learned intermediary") identified for this purpose and who have signed a DUA.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Started | 47 | 47
Completed | 41 | 37
Not Completed | 6 | 10
Not completed — Lost to Follow-up | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6) | 66 (7) | 66 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 44 | 39 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 39 | 42 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30 (3) | 31 (4) | 30 (4)
American Society of Anesthesiologists Status [Count of Participants; unit: Participants] — The grade is on a scale of 1-4 and is based on the patient's medical history, severity of known medical conditions, and current physical state to help predict if they can tolerate anesthesia and the conditions of surgery.
  Participants
    ASA 1 | 5 | 1 | 6
    ASA 2 | 39 | 46 | 85
    ASA 3 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (NRS, 0-10) With Ambulation on POD1
Description: The NRS (numeric rating scale) is a questionnaire that measures pain on a numeric scale, 0 (no pain) to 10 (worst pain imaginable). The questionnaire will be asked on post operative discharge day 1.
Time Frame: 24 hours Post Operative Discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
units on a scale | 4.55 (2.7) | 4.26 (3.03)
Statistical Analysis 1: Comparison: No PAI + ACB & IPACK vs PAI + ACB & IPACK; Test type: Non-Inferiority — Noninferiority Margin = (-Infinity, 1.28); p = 0.11, t-test, 1 sided

2. Secondary Outcome: Opioid Use (Cumulative Oral Morphine Equivalents POD0-POD2, 2 Weeks, 3 Months)
Description: Cumulative opioid consumption in morphine equivalents will be recorded post surgical discharge, 24h post surgical discharge, 48 hours post surgical discharge, 2 weeks post surgical discharge, and 3 months post surgical discharge.
Time Frame: post surgical discharge, 24 hours post surgical discharge, 48 hours post surgical discharge, 2 weeks post surgical discharge, and 3 months post surgical discharge.
Population: At post operative day 14 and 90, the number analyzed differ from the overall number because some subjects were lost to follow up.
Measure: Mean (Standard Deviation); unit: MME/day
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
MME/day
  post anesthesia care unit (PACU) | 25.45 (13.71) | 21.98 (12.02)
  post operative day (POD) 1 | 25.95 (20.04) | 22.16 (21.17)
  post operative day (POD) 2 | 37.3 (24.86) | 28.64 (30.21)
  post operative day (POD) 14: number analyzed (Participants) | 47 | 46
  post operative day (POD) 14 | 6.91 (10.53) | 6.68 (10.4)
  post operative day (POD) 90: number analyzed (Participants) | 41 | 37
  post operative day (POD) 90 | 0.27 (1.3) | 0.2 (1.23)
Statistical Analysis 1: Comparison: No PAI + ACB & IPACK vs PAI + ACB & IPACK; Test type: Non-Inferiority — a noninferiority margin of 1.0 and 10% attrition; p = 0.5, t-test, 2 sided — this is the calculated p-value; Mean Difference (Final Values) = .05

3. Secondary Outcome: NRS Pain With Movement
Description: The NRS (numeric rating scale) is a questionnaire that measures pain on a numeric scale, 0 (no pain) to 10 (worst pain imaginable). The questionnaire will focus on pain during movement and will be asked at pre-operation, in the post anesthesia care unit (PACU), at post operative (POD) 1, POD 2, and POD 3 months.
Time Frame: pre-operation, in the post anesthesia care unit (PACU), at post operative (POD) 1, POD 2, and POD 3 months
Population: the number of participants analyzed at POD 3 months is different due to lost to follow ups
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
units on a scale
  Pre-operation | 5.17 (2.52) | 5.85 (2.62)
  Post anesthesia care unit (PACU) | 5.7 (3.11) | 5.19 (2.92)
  Post operative day (POD) 1 | 4.55 (2.7) | 4.26 (3.03)
  Post operative day (POD) 2 | 6.68 (2.29) | 6.13 (2.62)
  Post operative day (POD) 3 months: number analyzed (Participants) | 41 | 37
  Post operative day (POD) 3 months | 1.02 (1.82) | 0.95 (1.47)

4. Secondary Outcome: Numerical Rating Scale (NRS) Pain Score at Rest
Description: The NRS (numeric rating scale) is a questionnaire that measures pain on a numeric scale, 0 (no pain) to 10 (worst pain imaginable). The questionnaire will focus on pain without movement involved and will be asked at pre-operation, post anesthesia care unit (PACU), post operative day (POD) 1, POD 2, and POD 3 months
Time Frame: from pre-operation, post anesthesia care unit (PACU), post operative day (POD) 1, POD 2, and POD 3 months
Population: number of participants analyzed at POD 3 months differed from overall number of participants due to lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
units on a scale
  pre-operation | 1.19 (2.05) | 1.79 (2.8)
  post anesthesia care unit (PACU) | 5.66 (3.17) | 5.06 (2.91)
  post operative day (POD) 1 | 2.36 (2.29) | 2.47 (2.86)
  post operative day (POD) 2 | 4.09 (2.95) | 4.13 (3.06)
  post operative day (POD) 3 months: number analyzed (Participants) | 41 | 37
  post operative day (POD) 3 months | 0.29 (0.93) | 0.46 (1.02)

5. Secondary Outcome: PAIN OUT Questionnaire at Preoperation
Description: The PAIN OUT questionnaire has multiple numeric scale questions on pain relief as well as pain intensity, along with Yes/No questions. There are also questions asking which pain relief techniques were used (multiple choice). All questions are scored on a scale of 0 to 10, with 0 meaning no pain/does not interfere/not at all and 10 meaning worst pain/completely interferes/extremely. A higher score means a worse outcome.
Time Frame: at preoperation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
score on a scale
  Least pain in 24 hours | 0.96 (1.96) | 1.45 (2.49)
  Worst pain in 24 hours | 6.57 (2.83) | 6.79 (2.7)
  Pain interfered or prevented you from activities in bed | 3.11 (3.51) | 3.02 (3.4)
  Pain interfered or prevented you from activities out of bed | 5.04 (3.55) | 5.94 (3.45)
  Pain interfered or prevented you from falling asleep | 2.49 (3.71) | 3.06 (4)
  Pain interfered or prevented you from staying asleep | 2.49 (3.71) | 3.06 (4)
  How much the pain caused you to feel anxious | 1.02 (2.55) | 1.89 (3.23)
  How much the pain caused you to feel depressed | 1.15 (2.66) | 1.6 (3.1)
  How much the pain caused you to feel frightened | 0.49 (1.72) | 1.02 (2.57)
  How much the pain caused you to feel helpless | 1.13 (2.68) | 1.02 (2.57)
  Severity of nausea | 0 (0) | 5 (0)
  Severity of drowsiness | 0 (0) | 0 (0)
  Severity of itching | 0 (0) | 0 (0)
  Severity of dizziness | 0 (0) | 0 (0)
  Were you allowed to participate in decisions about pain treatment? | 7.5 (5) | 10 (0)
  How satisfied are you with the results of your pain treatment? | 6.66 (5.77) | 10 (0)

6. Secondary Outcome: Quality of Recovery (POD1)
Description: Quality of Recovery (QoR-9), This questionnaire has three options for scale (not at all, some of the time, most of the time).
  The QoR-9 is a nine-item scale. Total QoR-9-scores range from 0 to 18, with higher scores indicating good recovery after anaesthesia.
  The questions focus on the overall well being of the patient. The questionnaire will be asked 24 hours post surgical discharge.
Time Frame: 24 hours post surgical discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
units on a scale | 16.62 (2.31) | 16.96 (2)

7. Secondary Outcome: Side Effects: Opioid-Related Symptom Distress Score (POD1)
Description: The Opioid-related symptom distress scale evaluates frequency, severity, bothersomeness for 12 symptoms. Each symptom is scored on a 4-point scale, with 0 meaning better outcome and 4 meaning worst outcome. The questionnaire will be asked 24 hours (POD 1) post surgical discharge.
Time Frame: 24 hours (POD 1) post surgical discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
score on a scale | .55 (.97) | .74 (1.09)

8. Secondary Outcome: Satisfaction With Pain Management (POD1)
Description: This questionnaire is a numeric scale from 0 (strongly dissatisfied) to 10 ( strongly satisfied). A higher number dictates a better outcome. This will be asked 24 hours post operative discharge.
Time Frame: 24 hours post operative discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
score on a scale | 9.7 (.81) | 9.66 (1.54)

9. Secondary Outcome: Blinding Assessment; Bang Question (POD1)
Description: There is no numeric scale for this questionnaire. It focuses on asking the subjects and the research assistant, which group they believe the subject were randomized to. This will be asked 24 hours post operative discharge.
Time Frame: 24 hours post operative discharge
Measure: Count of Participants; unit: Participants
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
Participants
  Subjects Guess: Guessed that the subject was in the "No PAI+ACB & IPACK" group | 10 | 8
  Subjects Guess: Guessed that the subject was in the "PAI+ACB & IPACK" group | 13 | 17
  Subjects Guess: Guessed "Don't know" | 24 | 22
  Research Assistant Guess: Guessed that the subject was in the "No PAI+ACB & IPACK" group | 0 | 3
  Research Assistant Guess: Guessed that the subject was in the "PAI+ACB & IPACK" group | 4 | 7
  Research Assistant Guess: Guessed "Don't know" | 43 | 37

10. Secondary Outcome: Douleur Neuropathique en 4 Questions (DN4) at Pre-operation, 3 Months
Description: The DN4 ( Douleur Neuropathique en 4 Questions) is a Yes/No questionnaire aimed at uncovering neuropathic pain symptoms. Each question is scored as yes or no, with yes = 1 point and no = 0 points. Total score is calculated by summing the total of the individual question scores, for a total score range of 0-10, with a score of greater than or equal to 4 indicating the patient may be suffering from neuropathic pain. The average score across all participants is calculated and reported for each time point.
Time Frame: Pre operative, 3 months post operative discharge.
Population: The number analyzed at POD 3 months differs from the overall number of participant due to lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
score on a scale
  at peroperation | 2.79 (1.35) | 2.62 (1.11)
  post operative day (POD) 3 months: number analyzed (Participants) | 41 | 37
  post operative day (POD) 3 months | 2.63 (.92) | 2.78 (.92)

11. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement
Description: The standard Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr.) questionnaire will be asked to evaluate orthopedic outcomes. The KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively.
  KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
  The questionnaire will be asked preoperatively, 6 weeks post operative discharge, 3 months post operative discharge.
Time Frame: preoperatively, 6 weeks post operative discharge, 3 months post operative discharge
Population: The number analyzed at 6 weeks and 3 months differ from the overall number due to lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
score on a scale
  at preoperation | 50.7 (16.2) | 49.61 (16.57)
  at 6 weeks: number analyzed (Participants) | 44 | 42
  at 6 weeks | 78.31 (11.36) | 77.05 (12.86)
  at 3 months: number analyzed (Participants) | 41 | 37
  at 3 months | 83.39 (13.83) | 83.60 (9.57)

12. Secondary Outcome: PAIN OUT Questionnaire at Post Operative Day (POD) 1
Description: as for outcome 5
Time Frame: at post operative day (POD) 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
score on a scale
  Least pain in 24 hours | 1.17 (2.05) | 1.34 (2.55)
  Worst pain in 24 hours | 6.53 (2.69) | 6.15 (2.97)
  Pain interfered or prevented you from activities in bed | 2.32 (3.85) | 2.4 (3.47)
  Pain interfered or prevented you from activities out of bed | 3.13 (3.85) | 2.4 (3.47)
  Pain interfered or prevented you from falling asleep | 1.06 (2.63) | .85 (2.29)
  Pain interfered or prevented you from staying asleep | 1.19 (2.84) | .96 (2.64)
  How much the pain caused you to feel anxious | .66 (2.1) | .23 (.94)
  How much the pain caused you to feel depressed | 0 (0) | .11 (.73)
  How much the pain caused you to feel frightened | .32 (1.62) | .26 (1.37)
  How much the pain caused you to feel helpless | .32 (1.62) | 0 (0)
  Severity of nausea | 6 (3.59) | 8.57 (2.9)
  Severity of drowsiness | 6.64 (2.69) | 6.72 (2.91)
  Severity of itching | 0 (0) | 2 (0)
  Severity of dizziness | 4.86 (3.23) | 6.1 (3.75)
  Were you allowed to participate in decisions about pain treatment? | 10 (0) | 9.76 (1.46)
  How satisfied are you with the results of your pain treatment? | 9.78 (.68) | 9.68 (1.53)

13. Secondary Outcome: PAIN OUT Questionnaire at Post Operative Day (POD) 14
Description: as for outcome 5
Time Frame: at post operative day (POD) 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 46
score on a scale
  Least pain in 24 hours | 1.72 (2.02) | 1.54 (2.11)
  Worst pain in 24 hours | 5.6 (2.62) | 5.26 (2.72)
  Pain interfered or prevented you from activities in bed | 2.68 (3.33) | 2.09 (2.98)
  Pain interfered or prevented you from activities out of bed | 1.81 (2.7) | 1.7 (2.46)
  Pain interfered or prevented you from falling asleep | 3.02 (3.92) | 2.85 (3.88)
  Pain interfered or prevented you from staying asleep | 3.15 (4.13) | 3.26 (3.96)
  How much the pain caused you to feel anxious | .66 (2.18) | .54 (1.86)
  How much the pain caused you to feel depressed | .38 (1.64) | .59 (1.83)
  How much the pain caused you to feel frightened | .09 (.58) | .07 (.44)
  How much the pain caused you to feel helpless | .23 (1.03) | .07 (.44)
  Severity of nausea | 5.5 (2.08) | 0 (0)
  Severity of drowsiness | 6 (4.58) | 4.4 (1.52)
  Severity of itching | 3.5 (.71) | 4.71 (2.81)
  Severity of dizziness | 0 (0) | 3 (0)
  Were you allowed to participate in decisions about pain treatment? | 9.76 (1.02) | 10 (0)
  How satisfied are you with the results of your pain treatment? | 9.61 (.89) | 9.71 (1.5)

14. Secondary Outcome: PAIN OUT Questionnaire at Post Operative Day (POD) 90
Description: as for outcome 5
Time Frame: at post operative day (POD) 90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 41 | 37
score on a scale
  Least pain in 24 hours | .05 (.22) | .24 (.86)
  Worst pain in 24 hours | 1.68 (2.18) | 1.81 (2.15)
  Pain interfered or prevented you from activities in bed | .29 (.98) | .89 (2.13)
  Pain interfered or prevented you from activities out of bed | .63 (1.39) | .65 (1.86)
  Pain interfered or prevented you from falling asleep | .61 (1.96) | .43 (1.48)
  Pain interfered or prevented you from staying asleep | .83 (2.06) | .86 (2.18)
  How much the pain caused you to feel anxious | .39 (1.39) | .35 (1.23)
  How much the pain caused you to feel depressed | .54 (2.01) | .27 (1.15)
  How much the pain caused you to feel frightened | 0 (0) | 0 (0)
  How much the pain caused you to feel helpless | 0 (0) | .14 (.82)
  Severity of nausea | 0 (0) | 0 (0)
  Severity of drowsiness | 3 (0) | 0 (0)
  Severity of itching | 7 (0) | 0 (0)
  Severity of dizziness | 0 (0) | 0 (0)
  Were you allowed to participate in decisions about pain treatment? | 9.51 (2.18) | 10 (0)
  How satisfied are you with the results of your pain treatment? | 9.48 (1.76) | 9.81 (.87)

15. Secondary Outcome: PAIN OUT Questionnaire at Preoperation / Percentage of Time in Severe Pain and Pain Relief
Description: The PAIN OUT questionnaire has multiple numeric scale questions on pain relief as well as pain intensity, along with Yes/No questions. There are also questions asking which pain relief techniques were used (multiple choice). All questions are scored on a scale of 0 to 10, with 0 meaning no pain/does not interfere/not at all and 10 meaning worst pain/completely interferes/extremely. A higher score means a worse outcome. This outcome records the percentage of time in severe pain and percentage pain relief, both scored from 0% to 100%.
Time Frame: at preoperation
Population: preoperative
Measure: Mean (Standard Deviation); unit: percentage of time or relief
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
percentage of time or relief
  Percentage of time in severe pain | 17.02 (22.83) | 18.09 (27.4)
  Pain relief in the first 24 hours | 5.5 (3.07) | 6.14 (2.91)

16. Secondary Outcome: PAIN OUT Questionnaire at Post Operative Day (POD) 1 / Percentage of Time in Severe Pain and Pain Relief
Description: as for outcome 15
Time Frame: at post operative day (POD) 1
Measure: Mean (Standard Deviation); unit: percentage of time or relief
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 47
percentage of time or relief
  the percentage of time in severe pain | 12.55 (22.98) | 11.49 (20.74)
  Pain relief in the first 24 hours | 9.93 (1.72) | 10.14 (1.85)

17. Secondary Outcome: PAIN OUT Questionnaire at Post Operative Day (POD) 14 / Percentage of Time in Severe Pain and Pain Relief
Description: as for outcome 15
Time Frame: at post operative day (POD) 14
Measure: Mean (Standard Deviation); unit: percentage of time or relief
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 47 | 46
percentage of time or relief
  The percentage of time in severe pain on a scale of 0 - 10 | 14.47 (25.44) | 17.61 (28.3)
  Pain relief in the first 24 hours on a scale of 0 - 10 | 9.65 (2.12) | 9.5 (2.53)

18. Secondary Outcome: PAIN OUT Questionnaire at Post Operative Day (POD) 90 / Percentage of Time in Severe Pain and Pain Relief
Description: as for outcome 15
Time Frame: at post operative day (POD) 90
Measure: Mean (Standard Deviation); unit: percentage of time or relief
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
Number analyzed (Participants) | 41 | 37
percentage of time or relief
  The percentage of time in severe pain | 9.02 (26.44) | 7.57 (23.5)
  Pain relief in the first 24 hours | 10.12 (2.63) | 10.37 (2.30)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from subject enrollment through completion of data collection (3 months after surgery).
Arm/Group | No PAI + ACB & IPACK | PAI + ACB & IPACK
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47 | 2/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No PAI + ACB & IPACK (N=47) | PAI + ACB & IPACK (N=47)
leakage at the incision site (Surgical and medical procedures) | 0 (0) | 1 (1)
postoperative myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
postoperative reduced range of motion (Surgical and medical procedures) | 0 (0) | 1 (1) — postoperative reduced range of motion requiring a knee manipulation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04749615/Prot_SAP_000.pdf